CLINICAL TRIAL: NCT00849654
Title: Phase I Dose-Escalation Study of Bruton's Tyrosine Kinase (Btk) Inhibitor PCI-32765 in Recurrent B Cell Lymphoma
Brief Title: Study of the Safety and Tolerability of PCI-32765 in Patients With Recurrent B Cell Lymphoma
Acronym: PCYC-04753
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pharmacyclics LLC. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PCYC-04753; NCT01177878 (obsolete NCT alias)
Record Dates: First submitted 2009-02-20; First posted 2009-02-24 (Estimated); Last update posted 2013-05-22 (Estimated); Status verified 2013-05

CONDITIONS: B-Cell Lymphoma; B-Cell Leukemia
Keywords: PCI-32765; Lymphoma; Lymphoma, Non-Hodgkin; Lymphoma, B-Cell; Burkitt Lymphoma; Lymphoma, B-Cell, Marginal Zone; Lymphoma, B-Cell, Diffuse; Lymphoma, Follicular; Lymphoma, Mantle Cell; Leukemia, Lymphoid; Leukemia, B-Cell; Waldenstrom macroglobulinemia; Bruton's Tyrosine Kinase
MeSH Terms: conditions — Lymphoma, B-Cell; Leukemia, B-Cell; Lymphoma; Lymphoma, Non-Hodgkin; Burkitt Lymphoma; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Leukemia, Lymphoid; Waldenstrom Macroglobulinemia | interventions — ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PCI-32765 (Experimental)
  Interventions: Drug: PCI-32765

INTERVENTIONS:
Drug: PCI-32765 — In the dose-escalation cohorts, PCI-32765 will be administered in 1.25, 2.5, 5.0, 8.3, 12.5, and 17.5 mg/kg/d dose orally once per day for 28 days followed by a 7-day rest period to determine the MTD. If MTD is not reached, dosing levels may be increased beyond 17.5mg/kg/d by 33% increments.
  In the continuous dosing cohorts, PCI-32765 will be administered in 8.3 mg/kg/day and 560 mg/day (fixed dose) dose orally once per day for 35 days.

SUMMARY:
The purpose of this study is to establish the safety and optimal dose of orally administered PCI-32765 in patients with recurrent B cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Women and men ≥ 18 years of age. There is no experience with this drug in a pediatric population.
* Body weight ≥ 40 kg.
* Recurrent surface immunoglobulin positive B cell non-Hodgkin's lymphoma (NHL) according to WHO classification, including small lymphocytic lymphoma/ chronic lymphocytic leukemia (SLL/CLL) lymphoplasmacytic lymphoma, including Waldenström's Macroglobulinemia (WM), and pre-identified DLBCL ABC subtype oFor the DLBCL-ABC cohort, documented, activated B-cell subtype by either immunohistochemistry or tissue microarray analysis.
* Measurable disease (for NHL, bidimensional disease ≥ 2 cm diameter in at least one dimension, for CLL ≥ 5000 leukemia cells/mm3, for WM presence of immunoglobulin M paraprotein with a minimum IgM level ≥ 1000 mg/dL and infiltration of bone marrow by lymphoplasmacytic cells), and pre-identified DLBCL ABC subtype by immunohistochemistry (IHC).
* Have failed ≥ 1 previous treatment for lymphoma and no standard therapy is available. Patients with diffuse large B cell lymphoma must have failed, refused or be ineligible for autologous stem cell transplant.
* ECOG performance status of ≤ 1.
* Ability to swallow oral capsules without difficulty.
* Willing and able to sign a written informed consent.

Exclusion Criteria:

* More than four prior systemic therapies (not counting maintenance rituximab), except for CLL patients. Salvage therapy/conditioning regimen leading up to autologous bone marrow transplantation is considered to be one regimen (This inclusion criterion does not apply to the DLBCL-ABC cohort).
* Prior allogeneic bone marrow transplant.
* Immunotherapy, chemotherapy, radiotherapy or experimental therapy within 4 weeks before first day of study drug dosing.
* Major surgery within 4 weeks before first day of study drug dosing.
* CNS involvement by lymphoma.
* Active opportunistic infection or treatment for opportunistic infection within 4 weeks before first day of study drug dosing.
* History of malabsorption.
* Laboratory abnormalities:

  * Creatinine > 1.5 × institutional upper limit of normal (ULN)
  * Total bilirubin > 1.5 x institutional ULN (unless elevated from documented Gilbert's syndrome)
  * AST or ALT > 2.5 × institutional ULN
  * Platelet count < 75,000/µL (unless patients have CLL and bone-marrow involvement, provided they are not transfusion-dependent)
  * Absolute neutrophil count (ANC) < 1500/µL (unless patients have CLL and bone-marrow involvement)
  * Hgb < 8.0 g/dL
* Uncontrolled illness including but not limited to: ongoing or active infection, symptomatic congestive heart failure (New York Heart Association Class III or IV heart failure), unstable angina pectoris, cardiac arrhythmia, and psychiatric illness that would limit compliance with study requirements.
* Risk factors for, or use of medications known to prolong QTc interval or that may be associated with Torsades de Pointes within 7 days of treatment start.
* QTc prolongation (defined as a QTc > 450 msecs) or other significant ECG abnormalities including 2nd degree AV block type II, 3rd degree AV block, or bradycardia (ventricular rate less than 50 beats/min). If the screening ECG has a QTc > 450 msecs, the ECG can be submitted for a centralized, cardiologic evaluation.
* History of myocardial infarction, acute coronary syndromes (including unstable angina), coronary angioplasty and/or stenting within the past 6 months.
* Known HIV infection.
* Hepatitis B sAg or Hepatitis C positive.
* Other medical or psychiatric illness or organ dysfunction which, in the opinion of the investigator, would either compromise the patient's safety or interfere with the evaluation of the safety of the study agent.
* Pregnant or lactating women (female patients of child-bearing potential must have a negative serum pregnancy test within 14 days of first day of drug dosing, or, if positive, a pregnancy ruled out by ultrasound).
* Women of child-bearing potential or sexually active men, unwilling to use adequate contraceptive protection during the course of the study.
* History of prior cancer < 2 years ago, except for basal cell or squamous cell carcinoma of the skin, cervical cancer in situ or other in situ carcinomas.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2009-02; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicity assessment for each patient. | At the end of the first 35 day cycle
Adverse events | 30 days after last dose of study drug
Pharmacokinetic/ Pharmacodynamic assessments | during Cycle 1

SECONDARY OUTCOMES:
Tumor response | at the end of Cycles 2, 4, and 6 unitl progression

CONTACTS AND LOCATIONS:
Overall Officials: Thorsten Graef, MD, PhD, Study Director — Pharmacyclics LLC.
Locations (9):
- United States (9):
  - Stanford University School of Medicine, Palo Alto, California
  - University of Chicago, Chicago, Illinois
  - National Cancer Institute, Bethesda, Maryland
  - New York Prebyterian Hospital Cornell Medical Center, New York, New York
  - Willamette Valley Cancer Institute/Research Ctr, Eugene, Oregon
  - University of Texas, MD Anderson, Houston, Texas
  - University of Vermont College of Medicine, Burlington, Vermont
  - Northwest Cancer Specialists, Vancouver Cancer Center, Vancouver, Washington
  - Yakima Valley Memorial Hospital/North Star Lodge Cancer Ctr, Yakima, Washington

REFERENCES:
- [Derived] Wilson WH, Young RM, Schmitz R, Yang Y, Pittaluga S, Wright G, Lih CJ, Williams PM, Shaffer AL, Gerecitano J, de Vos S, Goy A, Kenkre VP, Barr PM, Blum KA, Shustov A, Advani R, Fowler NH, Vose JM, Elstrom RL, Habermann TM, Barrientos JC, McGreivy J, Fardis M, Chang BY, Clow F, Munneke B, Moussa D, Beaupre DM, Staudt LM. Targeting B cell receptor signaling with ibrutinib in diffuse large B cell lymphoma. Nat Med. 2015 Aug;21(8):922-6. doi: 10.1038/nm.3884. Epub 2015 Jul 20. PMID 26193343
- [Derived] Marostica E, Sukbuntherng J, Loury D, de Jong J, de Trixhe XW, Vermeulen A, De Nicolao G, O'Brien S, Byrd JC, Advani R, McGreivy J, Poggesi I. Population pharmacokinetic model of ibrutinib, a Bruton tyrosine kinase inhibitor, in patients with B cell malignancies. Cancer Chemother Pharmacol. 2015 Jan;75(1):111-21. doi: 10.1007/s00280-014-2617-3. Epub 2014 Nov 8. PMID 25381051
- [Derived] Advani RH, Buggy JJ, Sharman JP, Smith SM, Boyd TE, Grant B, Kolibaba KS, Furman RR, Rodriguez S, Chang BY, Sukbuntherng J, Izumi R, Hamdy A, Hedrick E, Fowler NH. Bruton tyrosine kinase inhibitor ibrutinib (PCI-32765) has significant activity in patients with relapsed/refractory B-cell malignancies. J Clin Oncol. 2013 Jan 1;31(1):88-94. doi: 10.1200/JCO.2012.42.7906. Epub 2012 Oct 8. PMID 23045577
- See also: Related Info — http://www.pharmacyclics.com